CLINICAL TRIAL: NCT02806089
Title: Determinants of Muscle Strength in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UF9639
Record Dates: First submitted 2016-06-06; First posted 2016-06-20 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2017-01

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; malnutrition inflammation atherogenesis syndrome; muscle strength; muscle mass; lean body mass; physical activity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Muscle strength (Experimental): single evaluation (the day of inclusion) of muscle strength (by handheld dynamometer), muscle mass (by creatinine index estimation), lean body mass (by electrical bioimpedance analysis), physical activity (by "Voorrips" score questionnaire), inflammatory and nutritional status.
  Interventions: Device: Handheld dynamometer; Biological: Creatinine index; Device: Electrical bioimpedance analysis; Other: "Voorrips" score questionnaire; Biological: Inflammatory and nutritional status

INTERVENTIONS:
Device: Handheld dynamometer — Evaluation of muscle strength
Biological: Creatinine index — Evaluation of muscle mass using plasma creatinine level
Device: Electrical bioimpedance analysis — Evaluation of lean body mass
Other: "Voorrips" score questionnaire — Evaluation of physical activity
Biological: Inflammatory and nutritional status — Evaluation of C reactive protein and albumin

SUMMARY:
Aim of this study is to determine in chronic kidney disease patients:

* the involvement of malnutrition inflammation and atherogenesis syndrome (increase in C reactive protein and decrease in serum albumin) on voluntary muscle strength impairment
* the relationship between voluntary muscle strength and muscle mass
* the relationship between voluntary muscle strength and lean body mass
* the correlation between voluntary muscle strength and physical activity

DETAILED DESCRIPTION:
Aim of this study is to determine in chronic kidney disease patients:

* the involvement of malnutrition inflammation and atherogenesis syndrome (increase in C reactive protein and decrease in serum albumin) on voluntary muscle strength impairment (estimated by handheld dynamometer)
* the relationship between voluntary muscle strength and muscle mass (estimated by creatinine index)
* the relationship between voluntary muscle strength and lean body mass (estimated by bioelectrical impedance analysis)
* the correlation between voluntary muscle strength and physical activity (the physical activity being estimated by the "Voorrips" score questionnaire)

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease patient with extrarenal replacement therapy by hemodialysis for at least 3 months
* stable clinical condition (absence of infection, stroke or acute decompensation)

Exclusion Criteria:

* chronic kidney disease without extrarenal replacement therapy
* history of renal transplantation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Voluntary muscle strength evaluated by handheld dynamometer | 1 day
  data will be measured in Newton.meter

SECONDARY OUTCOMES:
Muscle mass estimated by creatinine index evaluation | 1 day
  data will be obtained from plasma creatinine level and will be expressed in milligram/kilogram/day)
Lean body mass evaluated by electrical bioimpedance analysis | 1 day
  data will be expressed in kilogram
Physical activity estimated using the "Voorrips" score questionnaire | 1 day
  the score represents the daily physical activity according to a validated scale
C reactive protein level | 1 day
  the parameter will be measured in milligram/liter
Albumin level | 1 day
  the parameter will be measured in gram/liter

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul CRISTOL, Prof, Principal Investigator — CHU Lapeyronie, Department of Biochemistry and Hormonology, Montpellier, FRANCE
Locations (3):
- France (3):
  - AIDER, Montpellier
  - GCS Help Lapeyronie, CHU Montpellier, Montpellier
  - AIDER, Nîmes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Souweine JS, Kuster N, Chenine L, Rodriguez A, Patrier L, Morena M, Badia E, Chalabi L, Raynal N, Ohresser I, Leray-Moragues H, Mercier J, Hayot M, Le Quintrec M, Gouzi F, Cristol JP. Physical inactivity and protein energy wasting play independent roles in muscle weakness in maintenance haemodialysis patients. PLoS One. 2018 Aug 1;13(8):e0200061. doi: 10.1371/journal.pone.0200061. eCollection 2018. PMID 30067754